CLINICAL TRIAL: NCT01307475
Title: Freeman-Sheldon Syndrome Quality of Life Study (FSS-QLS): Cross-sectional Study of Concomitant Disorder-Specific Contributors to Quality of Life and Clinical Outcome
Brief Title: Study of Quality of Life in Freeman-Sheldon Syndrome and Related Conditions
Acronym: FSS-QLS
Status: Terminated | Type: Observational
Why Stopped: Most study procedures incorporated into NCT01144741, some in NCT01306994
Sponsor: Freeman-Sheldon Research Group, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 000082; U1111-1120-5996 (Other: World Health Organisation, Universal Trial Number)
Record Dates: First submitted 2011-02-27; First posted 2011-03-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Arthrogryposis; Craniofacial Abnormalities; Posttraumatic Stress Disorder; Depressive Disorder
Keywords: Chronic Post-Traumatic Stress Disorder; Delayed Onset Post-Traumatic Stress Disorder; Post-Traumatic Neuroses; Posttraumatic Neuroses; Post-Traumatic Stress Disorders; Posttraumatic Stress Disorders; PTSD; Post TraumaticStress Disorder; Endogenous Depression; Neurotic Depression; Depressive Syndrome; Melancholia; Depressive Neurosis; Unipolar Depression; Depressive Symptoms; Emotional Depression; Quality of Life
MeSH Terms: conditions — Arthrogryposis; Craniofacial Abnormalities; Stress Disorders, Post-Traumatic; Depressive Disorder; Depression | interventions — Multicenter Studies as Topic; Health Records, Personal; Restraint, Physical; Independent Medical Evaluation; Psychometrics; Lactic Acid; Glucose; Hematologic Tests; Adenosine Triphosphate; Glucose Tolerance Test; Blood Glucose

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood samples will be taken but no retention is expected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Proband Group: Patients identified with FSS or a related condition
  Interventions: Other: PTSD Checklist-Specific; Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale; Other: Functional Enquiry Form; Other: Strength, Joint ROM, Girth and Length Measurements; Other: Study Physical Examination; Other: PTSD, Depression, and FSS-Focused Examination; Other: Freeman-Sheldon Specific Quality of Life Survey; Other: Lactate, Glucose, and Adenosine Triphosphate Blood Levels
- Family Group: Persons who are genetically or legally related to a person with FSS or related condition
  Interventions: Other: PTSD Checklist-Specific; Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale; Other: Functional Enquiry Form; Other: Strength, Joint ROM, Girth and Length Measurements; Other: Study Physical Examination; Other: PTSD, Depression, and FSS-Focused Examination; Other: Freeman-Sheldon Specific Quality of Life Survey; Other: Lactate, Glucose, and Adenosine Triphosphate Blood Levels
- Other Affected Individuals Group: Persons who have had significant and meaningful contact with a person with FSS or related condition but do not qualify for family group enrolment
  Interventions: Other: PTSD Checklist-Specific; Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale; Other: Functional Enquiry Form; Other: Strength, Joint ROM, Girth and Length Measurements; Other: Study Physical Examination; Other: PTSD, Depression, and FSS-Focused Examination; Other: Freeman-Sheldon Specific Quality of Life Survey; Other: Lactate, Glucose, and Adenosine Triphosphate Blood Levels

INTERVENTIONS:
Other: PTSD Checklist-Specific — Completed by patients before clinical examination; it is a 17-item survey listing of symptoms of posttraumatic stress disorder.
  Other Names: PCL-S; PCL-C; PTSD Checklist-Civilian
Other: Modified Flanagan Quality of Life Scale — Completed by patients before clinical examination; it is a 16-item survey designed for use in persons with chronic illness.
  Other Names: QOLS; Flanagan Quality of Life Scale; Quality of Life Scale
Other: Center for Epidemiologic Studies Depression Scale — Completed by patients before clinical examination; it is a 20-item survey that asks about depressive feelings and behaviours in the past week.
  Other Names: CES-D
Other: Functional Enquiry Form — Completed by patients before clinical examination; it is a checklist of medical problems.
  Other Names: FSRG Form 08; health history; review of systems; systems review; medical history; personal health history
Other: Strength, Joint ROM, Girth and Length Measurements — Completed during the clinical examination by the researchers, it is a structured approach to evaluation of muscles, joints, arms, thighs, and legs.
  Other Names: SF 527; Standard Form 527; musculoskeletal examination; musculoskeletal exam; musculoskeletal evaluation; musculoskeletal assessment; extremity examination; extremity evaluation; extremity assessment; extremity exam
Other: Study Physical Examination — Completed during the clinical examination by the researchers, it is a structured approach to a full physical examination, minus breasts, genitalia or rectum.
  Other Names: FSRG Form 14; physical examination; physical evaluation; physical assessment; medical examination; medical evaluation; medical assessment; full medical examination; full medical evaluation; full medical assessment; periodic medical examination; periodic medical evaluation; periodic medical assessment; annual medical examination; annual medical evaluation; annual medical assessment; yearly medical examination; yearly medical evaluation; yearly medical assessment; full physical examination; full physical evaluation; full physical assessment; complete physical examination; complete physical evaluation; complete physical assessment; yearly physical examination; yearly physical evaluation; yearly physical assessment; annual physical examination; annual physical evaluation; annual physical assessment; periodic physical examination; periodic physical evaluation; periodic physical assessment; screening physical examination; screening physical evaluation; screening physical assessment; screening physical; physical; periodic physical; annual physical; annual check-up; annual check up; yearly physical; yearly check up; yearly check-up; check up; check-up; medical check-up; medical check up; annual medical check-up; annual medical check up; yearly medical check-up; yearly medical check up; periodic medical check-up; periodic medical check up; periodic health evaluation; periodic health assessment; annual health evaluation; annual health assessment; yearly health evaluation; yearly health assessment; screening health evaluation; screening health assessment; screening medical examination; screening medical evaluation; screening medical assessment; med check
Other: PTSD, Depression, and FSS-Focused Examination — Completed during the clinical examination by the researchers, it is a structured approach to evaluation of symptoms, signs, and perceptions that may be related to FSS, PTSS, or depressive problems.
  Other Names: psychiatric examination; psychiatric evaluation; psychiatric assessment; diagnostic mental health examination; diagnostic mental health evaluation; diagnostic mental health assessment; diagnostic psychiatric examination; diagnostic psychiatric evaluation; diagnostic psychiatric assessment; intake examination; intake evaluation; intake assessment; mental health evaluation; mental health examination; mental health assessment; psychological examination; psychological evaluation; psychological assessment; psychological intake examination; psychological intake evaluation; psychological intake assessment; PTSD examination; PTSD evaluation; PTSD assessment; posttraumatic stress disorder evaluation; posttraumatic stress disorder examination; posttraumatic stress disorder assessment; post-traumatic stress disorder evaluation; post-traumatic stress disorder examination; post-traumatic stress disorder assessment; post traumatic stress disorder evaluation; post traumatic stress disorder examination; post traumatic stress disorder assessment; depression diagnostic examination; depression diagnostic evaluation; depression diagnostic assessment; depression evaluation; depression assessment
Other: Freeman-Sheldon Specific Quality of Life Survey — Completed after data analysis from the existing surveys and clinical examination, it will be a specific quality of life survey developed and tested during the study; it will take into consideration individual's total health outcome.
  Other Names: psychometric test development; psychometric testing; psychometric test validation; quality of life scale development; quality of life scale validation; quality of life survey development; quality of life survey validation; quality of life measure development; quality of life measure validation
Other: Lactate, Glucose, and Adenosine Triphosphate Blood Levels — Completed during the clinical examination by the researchers, lactate, glucose, and free and total adenosine triphosphate blood levels are determined at rest.
  Other Names: ATP levels; ATP blood levels; adenosine triphosphate test; blood test for ATP; blood test for adenosine triphosphate; ATP blood test; adenosine triphosphate blood test; ATP test; glucose test; glucose blood test; sugar test; lactic acid levels; lactic acid blood test; lactate blood test; lactate levels

SUMMARY:
Freeman-Sheldon syndrome (FSS) is a rare human neuromusculoskeletal disorder present before birth, involving primarily limb and craniofacial deformities.

The hypotheses in the present study of FSS and related conditions are: (1) FSS and related conditions are associated with higher rates of posttraumatic stress symptoms (PTSS), depression, and reduced quality of life than is observed in the general population; (2) persons close to an individual with FSS or related condition suffer similarly; and (3) current measures, which are single-disease specific (i.e., PTSS, depression, craniofacial deformities, or limb deformities), do not capture the unique picture of FSS and related conditions, which involve both limb and craniofacial deformities in an intellectually capable individual.

There have been no studies looking at quality of life associated with FSS. Some authors have looked at quality of life in persons with facial differences; other authors have looked at bone and joint problems. Many other authors have looked at PTSS and depression caused by health problems and bad medical experiences. No authors have looked at these problems when they happen together, as they do in FSS. Because of the above, there may be differences in patients that have FSS versus patients in previous quality of life studies. The study will also develop and validate an outcomes-based quality of life survey for FSS and related conditions.

DETAILED DESCRIPTION:
This study is a research project initiated by the graduate research student (Mikaela I. Poling) and assisted by the clinical genetics fellow and graduate student (Andrés Morales) in partial fulfilment the requirements for their Masters degrees in Clinical and Applied Physiology, under approval, direction, and supervision of the study PI (Rodger J. McCormick).

Mental Health and Congenital Deformities:

Apajasalo et al. (1998) found significantly decreased health-related quality of life versus controls among adults and youth ages with chondrodysplasias. Differences in adult scores were in the areas of mobility, usual activities, and sexual activity and discomfort. Youth scores differed more in school and hobbies and friends and physical appearance. Didierjean-Pillet (2002) stressed concern for aesthetics of reconstruction in consideration of psychiatric impacts of congenital deformities in psychosocial functioning. Nagata et al. (2008) found that 20% of mothers with children operated on for congenital disease were likely to have post-traumatic stress disorder (PTSD). They found that pro-active, effective participation in the child's care may alleviate PTSS. Vitale et al. (2005) found quality of life survey scores among clubfoot patients compatible with age-matched controls, in agreement with Roye (2001), and not correlated to radiograph appearance. They advised quality of life survey scores be primary endpoint in determining therapeutic outcome. Engell et al. (2007) found significant post-operative improvement in the Short Form-12 Health Survey physical component scale in congenital clubbed-foot patients in the Danish Twin Registry. Vitale et al. (2001) observed that tailored quality of life scales were required for paediatric orthopaedic populations. Hawkins and Radcliffe (2006) concluded there was a lack of appropriate and validated PTSD measures for paediatric patients. Part of this problem of lacking validated paediatric PTSD measures was likely do to non-comprehensive Diagnostic and Statistical Manual of Mental Disorders IV Text-Revision criteria.

Relevance to Current Study:

Because FSS-related deformities were more comprehensive, treatment-resistant, and associated with poorer clinical outcome, quality of life studies not including a subset of FSS patients may not be appropriate in the more challenging clinical picture of FSS-related deformities. In many conditions, disorder-specific quality of life measures (QLM) showed increased sensitivity and specificity over general QLMs and were important therapeutic tools to assess efficacy of and prioritise interventions. Results of disorder-specific QLMs were important predictors of clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Freeman-Sheldon syndrome,
* Sheldon-Hall syndrome,
* Distal arthrogryposis type 1, or
* distal arthrogryposis type 3
* Deceased probands with enough clinical information available to satisfy study requirements
* Probands who participated in a prior Freeman-Sheldon Research Group (FSRG)-study are automatically accepted, since their diagnoses have been confirmed by FSRG clinical faculty.
* Probands with a reported qualifying diagnosis, who have not participated in a prior FSRG-study, will be required to complete the complete a survey from a prior study and provide photographs and any requested medical records to confirm their diagnoses.
* Family members and other close contacts may enrol, so long as they have either resided with or had substantial and prolonged contact with a proband, who has an FSRG-verified qualifying diagnosis. Investigators will make the final decision on a case-by-case basis, based on information provided.

Exclusion Criteria:

* Patients with other anomalies, not having one of the above syndromes, will not be accepted.
* Deceased probands will not be accepted for analysis, without enough clinical data available to satisfy study data collection requirements.
* Patients or parents of minor children not willing to give consent will not be included.
* Family members or other contacts that neither resided with nor had substantial and prolonged contact with the proband.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients, family, and others affected world-wide are welcome, so long as they currently or previously have had significant and meaningful contact with a person who has a qualifying diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-02; Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Situational Mental Health in Persons with FSS or Related Condition | Evaluated during 1-2 study visits (lasting an average of 1-3 hours each) and in self-completed surveys, over an average of 2-4 years from enrolment
  Increased frequency of mental health symptoms and diagnoses (PTSS, Depression, and reduced quality of life) over expected for general population

SECONDARY OUTCOMES:
Situational Mental Health in Family and Others with a Close Relationship to a Person with FSS or Related Condition | Evaluated during 1-2 study visits (lasting an average of 1-3 hours each) and in self-completed surveys, over an average of 2-4 years from enrolment
  Increased frequency of mental health symptoms and diagnoses (PTSS, Depression, and reduced quality of life) over expected for general population
Current Survey Correlation with Disorder-Specific Survey for FSS and Related Conditions | Evaluated during 1-2 study visits (lasting an average of 1-3 hours each) and in self-completed surveys, over an average of 2-4 years from enrolment
  Ability of current surveys to capture full picture of quality of life for persons, families, and others affected by FSS and related conditions will be assessed to determine need for a disorder-specific survey and usefulness of existing surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Chamberlain, MD, Principal Investigator — Freeman-Sheldon Research Group, Inc.
Locations (2):
- Freeman-Sheldon Research Group, Inc. Headquarters, Buckhannon, West Virginia, United States
- San Juan de Dios General Hospital, Guatemala City, Guatemala

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared, due to concerns involved in masking identities of individuals with such a rare condition.

REFERENCES:
- [Background] Apajasalo M, Sintonen H, Rautonen J, Kaitila I. Health-related quality of life of patients with genetic skeletal dysplasias. Eur J Pediatr. 1998 Feb;157(2):114-21. doi: 10.1007/s004310050781. PMID 9504784
- [Background] Didierjean-Pillet A. [Psychological approach to congenital hand deformities. Congenital deformities, the desire to know]. Ann Chir Plast Esthet. 2002 Feb;47(1):2-8. doi: 10.1016/s0294-1260(01)00079-6. French. PMID 11980349
- [Background] Nagata S, Funakosi S, Amae S, Yoshida S, Ambo H, Kudo A, Yokota A, Ueno T, Matsuoka H, Hayashi Y. Posttraumatic stress disorder in mothers of children who have undergone surgery for congenital disease at a pediatric surgery department. J Pediatr Surg. 2008 Aug;43(8):1480-6. doi: 10.1016/j.jpedsurg.2007.12.055. PMID 18675639
- [Background] Vitale MG, Choe JC, Vitale MA, Lee FY, Hyman JE, Roye DP Jr. Patient-based outcomes following clubfoot surgery: a 16-year follow-up study. J Pediatr Orthop. 2005 Jul-Aug;25(4):533-8. doi: 10.1097/01.bpo.0000157999.38424.ba. PMID 15958910
- [Background] Roye BD, Vitale MG, Gelijns AC, Roye DP Jr. Patient-based outcomes after clubfoot surgery. J Pediatr Orthop. 2001 Jan-Feb;21(1):42-9. doi: 10.1097/00004694-200101000-00010. PMID 11176352
- [Background] Vitale MG, Levy DE, Johnson MG, Gelijns AC, Moskowitz AJ, Roye BP, Verdisco L, Roye DP Jr. Assessment of quality of life in adolescent patients with orthopaedic problems: are adult measures appropriate? J Pediatr Orthop. 2001 Sep-Oct;21(5):622-8. PMID 11521031
- [Background] Hawkins SS, Radcliffe J. Current measures of PTSD for children and adolescents. J Pediatr Psychol. 2006 May;31(4):420-30. doi: 10.1093/jpepsy/jsj039. Epub 2005 Jun 9. PMID 15947119
- [Result] McCormick RJ, Poling MI, Portillo AL, Chamberlain RL. Preliminary experience with delayed non-operative therapy of multiple hand and wrist contractures in a woman with Freeman-Sheldon syndrome, at ages 24 and 28 years. BMJ Case Rep. 2015 Jul 14;2015:bcr2015210935. doi: 10.1136/bcr-2015-210935. PMID 26174733
- [Result] McCormick RJ, Poling MI, Chamberlain RL. Bilateral patellar tendon-bearing Symes-type prostheses in a severe case of Freeman-Sheldon syndrome in a 21-year-old woman presenting with uncorrectable equinovarus. BMJ Case Rep. 2015 Jul 15;2015:bcr2015211338. doi: 10.1136/bcr-2015-211338. PMID 26178231
- [Result] Chamberlain RL, Poling MI, Portillo AL, Morales A, Ramirez RR, McCormick RJ. Freeman-Sheldon syndrome in a 29-year-old woman presenting with rare and previously undescribed features. BMJ Case Rep. 2015 Oct 22;2015:bcr2015212607. doi: 10.1136/bcr-2015-212607. PMID 26494722
- [Result] Poling MI, Dufresne CR, Chamberlain RL. Dr Ben Franklin and an unusual modern-day cure for recurrent pleuritis. Br J Gen Pract. 2017 Jan;67(654):32-33. doi: 10.3399/bjgp17X688705. No abstract available. PMID 28034943
- [Result] Poling MI, Morales Corado JA, Chamberlain RL. Findings, phenotypes, and outcomes in Freeman-Sheldon and Sheldon-Hall syndromes and distal arthrogryposis types 1 and 3: protocol for systematic review and patient-level data meta-analysis. Syst Rev. 2017 Mar 6;6(1):46. doi: 10.1186/s13643-017-0444-4. PMID 28264711